CLINICAL TRIAL: NCT05876572
Title: A Pharmacokinetic/Pharmacodynamic (PK/PD) Evaluation of Naloxone Following Intradermal Injection in Humans
Brief Title: Blood Naloxone Levels Following Intradermal Injection in Humans
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Currently does not have active IRB status
Sponsor: Johns Hopkins University (Other)
Collaborators: DEKA S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00380585
Record Dates: First submitted 2023-05-10; First posted 2023-05-25 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Opioid Overdose
Keywords: naloxone; pharmacokinetics; pharmacodynamics; intradermal; Opioid receptor
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- healthy volunteer adults (Other)
  Interventions: Drug: intradermal naloxone; Device: microneedle injection

INTERVENTIONS:
Drug: intradermal naloxone — One time 8 mg/0.1 mL dose of naloxone to be administered intradermally
Device: microneedle injection — Intradermal delivery of naloxone using microneedle

SUMMARY:
The main purpose of this study is to evaluate pharmacokinetics/pharmacodynamics of intradermal administration of naloxone in healthy adult subjects.

DETAILED DESCRIPTION:
Using approved drug formulations, injection devices, and assays, the investigators seek to determine the pharmacokinetics and pharmacodynamics of naloxone in human subjects using an intradermal delivery route. The long-term goal is to develop a product with better pharmacokinetic (PK) and pharmacodynamic (PD) properties than current delivery systems used in opioid overdose rescue. To the best of the investigators knowledge, this is the first study administering naloxone via an intradermal route in humans. Using an FDA-approved intranasal drug formulation, the investigators will administer 8mg/0.1ml of naloxone into the highly vascular dermal layer of the skin using microneedles in 3 healthy volunteer participants and measure plasma concentrations of naloxone for 60 minutes after injection. The investigators primary outcome measure is detectable levels of naloxone in plasma. Secondary outcome measures will be estimates of PK values derived from time versus concentration data.

ELIGIBILITY:
Inclusion Criteria:

* Ability to participate in the informed consent process
* Good peripheral venous access for proposed pharmacokinetic sampling
* Has not taken an investigational drug within prior 30 days (or 5 half-lives, whichever is longer)

Exclusion Criteria:

* Allergy to Naloxone or vehicle constituents (namely parabens)
* Active substance use as defined by a positive screen for drugs of abuse within seven days of study participation
* History of substance use disorder
* Taking opiate/opioid medications for any indication
* Chronic pain disorder
* Pregnant or breastfeeding
* Adults lacking capacity to consent, non-English speaking persons, or prisoners.
* Other medical history or active conditions deemed not safe for participation by the investigator
* Hematocrit <35%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Detection of Plasma Naloxone Concentration (ng/mL) using High Performance Liquid Chromatography/Tandem Mass Spectrometry (HPLC-MS/MS). | up to 60 minutes
  Plasma Naloxone concentration (ng/mL) will be measured using HPLC-MS/MS at multiple timepoints following an intradermal injection of 8mg dose of Naloxone. The primary outcome is the presence or absence of detectable Naloxone at any time point. Time points include T0 (pre-Naloxone), 1, 2, 4, 6, 8, 12.5, 15, 30, 45, and 60 minutes after Naloxone treatment. Multiples of time points between participants will be taken as a simple mean average for that specific time point, and any samples below the limit of assay detection will be excluded from calculation.

SECONDARY OUTCOMES:
Measurement of the maximum plasma concentration (Cmax; ng/mL) of Naloxone using HPLC-MS/MS following a single 8mg dose of intradermally delivered Naloxone. | up to 60 minutes
  Using the data collected for the primary outcome, a secondary analysis will be done to determine the maximum concentration of Naloxone (Cmax) reached in plasma during the course of 60 minutes after an intradermal injection of Naloxone. Cmax will be taken as the highest mean average concentration (ng/ml) of plasma naloxone achieved at any given time point (times listed under primary outcomes). In conjunction with other data from this study, absorption rate and other important pharmacologic measures can be estimated to guide development of future phase 1 pharmacokinetic trials.
Assessment of the time (minutes) at which the maximum Naloxone concentration (ng/mL) is detected in plasma (Tmax) by HPLC-MS/MS after a single 8mg dose of intradermally delivered Naloxone. | up to 60 minutes
  Using the data collected for the primary outcome, another secondary analysis will be done to determine the time at which Naloxone concentration reaches a maximum during the course of 60 minutes after an intradermal injection of Naloxone. This will be determined by selecting the time point at which the highest mean average concentration (ng/ml) of plasma Naloxone is achieved among any of the times point listed under primary outcomes. In conjunction with other data from this study, absorption rate and other important pharmacologic measures can be estimated to guide development of future phase 1 pharmacokinetic trials.
Assessment of Naloxone exposure (mg*h/L) over 60 minutes (AUC 0-60) as measured by HPLC-MS/MS of plasma samples collected after a single 8mg dose of intradermally delivered Naloxone. | up to 60 minutes
  Additionally, Naloxone concentrations (ng/mL) taken from the above experiment will be averaged (mean) for each time point and then used to calculate the Area Under the Curve (AUC; mg*h/L) as a measure of Naloxone exposure over the course of 60 minutes after intradermal Naloxone injection. In conjunction with other data from this study, absorption rate and other important pharmacologic measures can be estimated to guide development of future phase 1 pharmacokinetic trials.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Rosenblatt, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No